CLINICAL TRIAL: NCT05280470
Title: A Phase 2, Multicenter, Randomized, Open-label Study of Ifinatamab Deruxtecan (I-DXd), a B7-H3 Antibody Drug Conjugate (ADC), in Subjects With Pretreated Extensive-stage Small Cell Lung Cancer (ES-SCLC) (IDeate-Lung01)
Brief Title: Ifinatamab Deruxtecan (I-DXd) in Subjects With Pretreated Extensive-Stage Small Cell Lung Cancer (ES-SCLC)
Acronym: IDeate-Lung01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS7300-127; 2022-000503-13 (EudraCT Number); 2041220019 (Other: jRCT)
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Extensive-stage Small-cell Lung Cancer
Keywords: Relapsed/Refractory Extensive-stage Small-cell Lung Cancer; DS-7300a; B7-H3 Antibody Drug Conjugate; Ifinatamab Deruxtecan; I-DXd
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ifinatamab Deruxtecan (8 mg/kg) (Experimental): Participants will be randomized to receive I-DXd at 8 mg/kg.
  Interventions: Drug: Ifinatamab Deruxtecan (I-DXd)
- Ifinatamab Deruxtecan (12 mg/kg) (Experimental): Participants will be randomized to receive I-DXd at 12 mg/kg.
  In Part 2, all participants will receive I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab Deruxtecan (I-DXd)

INTERVENTIONS:
Drug: Ifinatamab Deruxtecan (I-DXd) — I-DXd will be administered as an intravenous (IV) infusion on Day 1 of each 21-day cycle (every Q3W).
  Other Names: DS-7300a

SUMMARY:
This 2-part study intends to define the recommended Phase 2 dose of ifinatamab deruxtecan (I-DXd) based on the efficacy, safety, and pharmacokinetics (PK) results observed in participants with Extensive-stage Small Cell Lung Cancer (ES-SCLC) who received at least 1 prior line of platinum-based chemotherapy and a maximum of 3 prior lines of therapy (Part 1) and a minimum of two previous lines of systemic therapy (Part 2). This study will also investigate I-DXd anti-tumor activity in this population.

DETAILED DESCRIPTION:
This study will consist of 2 parts: dose optimization (Part 1) and extension (Part 2). In the dose optimization part of the study (Part 1), approximately 80 participants with at least 1 prior line of platinum-based chemotherapy and a maximum of 3 prior lines of therapy will be enrolled. Two I-DXd doses will be tested (8 mg/kg Q3W and 12 mg/kg Q3W). In the extension part of the study (Part 2), approximately 70 participants with a minimum of two previous lines of systemic therapy will be enrolled. I-DXd will be administered at the selected dose of 12 mg/kg Q3W.

In Part 1, eligible participants will be randomized in a 1:1 ratio to receive one of the two dose levels of I-DXd. Randomization will be stratified by:

1. Prior receipt or of an anti-programmed death-ligand 1 (PD-[L]1) antibody (yes/no)
2. The chemotherapy-free interval (CTFI) from completion of the first-line therapy to the date of documented radiological Progressive Disease of <90 days vs. ≥90 days in second-line participants as well as the number of lines of therapy. Thus, the stratification factor includes three categories: (1) second-line participants with CTFI <90 days, (2) second-line participants with CTFI ≥90 days, and (3) third- and fourth-line participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible for enrollment into the study:

* Sign and date the informed consent form (ICF) prior to the start of any study-specific qualification procedures.
* Participant must have at least one lesion, not previously irradiated, amenable to core biopsy.
* Male or female subjects aged ≥18 years (follow local regulatory requirements if the legal age of consent for study participation is >18 years old).
* Histologically or cytologically documented ES-SCLC.
* At least one measurable lesion according to RECIST v1.1 as assessed by the investigator.
* Prior therapy with at least one platinum-based line as systemic therapy for extensive-stage disease with at least two cycles of therapy (except in the case of early objective PD) and beginning with protocol version 3.0, a minimum of two previous lines of systemic therapy.
* Documentation of radiological disease progression on or after most recent systemic therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.

Exclusion Criteria:

Participants who meet any of the following criteria will be disqualified from entering the study:

* Prior treatment with orlotamab, enoblituzumab, or other B7-H3 targeted agents, including I-DXd.
* Prior discontinuation of an antibody drug conjugate (ADC) that consists of an exatecan derivative (eg, trastuzumab deruxtecan) due to treatment-related toxicities.
* Clinically active brain metastases, spinal cord compression or leptomeningeal carcinomatosis, defined as untreated or symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms.
* Any of the following conditions within the past 6 months: cerebrovascular accident, transient ischemic attack, or another arterial thromboembolic event.
* Clinically significant corneal disease.
* Uncontrolled or significant cardiovascular disease.
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required corticosteroids, current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses,
* Chronic steroid treatment (dose of 10 mg daily or more prednisone equivalent), except for low-dose inhaled steroids (for asthma/COPD) or topical steroids (for mild skin conditions) or intra-articular steroid injections.
* History of malignancy other than SCLC within the 3 years prior to enrollment, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, superficial gastrointestinal (GI) tract tumors and non-muscle invasive bladder cancer curatively resected by endoscopic surgery.
* History of allogeneic bone marrow, stem cell, or solid organ transplant.
* Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute- Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE V5.0), Grade ≤1 or baseline.
* History of hypersensitivity to the drug substances, inactive ingredients in the drug product or severe hypersensitivity reactions to other monoclonal antibodies.
* Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection.
* Has active or uncontrolled hepatitis B or C infection.
* Active, known, or suspected autoimmune disease.
* Any evidence of severe or uncontrolled systemic diseases (including active bleeding diatheses, psychiatric illness/social situations, substance abuse).
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Female who is pregnant or breast-feeding or intends to become pregnant during the study.
* Prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the participant.
* Known human immunodeficiency virus (HIV) infection that is not well controlled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Objective Response Rate (ORR) Based on Blinded Independent Central Review (BICR) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | Up to approximately 36 months
  ORR was defined as the percentage of participants who achieved a best overall response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), assessed by BICR based on RECIST version 1.1. For all target, non-target, and new lesions, CR was defined as a disappearance of all lesions and PR was defined as at least a 30% decrease in the sum of diameters of all lesions.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | Up to approximately 36 months
  TEAEs are defined as new adverse events (AEs) that occur after the dose of study drug or as AEs that were present prior to the dose of study drug but which worsened in severity after the start of study drug.
Progression-Free Survival (PFS) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | From enrollment until disease progression or death (whichever occurs first), up to approximately 36 months
  PFS is defined as the time interval from the date of enrollment to the date of disease progression based on RECIST v1.1 or death due to any cause. PFS will be assessed by BICR and investigator.
Duration of Response (DoR) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | From enrollment until disease progression or death (whichever occurs first), up to approximately 36 months
  DoR is defined as the time from the date of first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression based on RECIST v1.1 or to death due to any cause, whichever occurs first. DoR will be assessed by BICR and investigator.
Overall Survival (OS) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | From enrollment until death, up to approximately 36 months
  OS is defined as the time interval from the date of enrollment to the date of death due to any cause or last contact follow-up, whichever occurs first.
Time to Response (TTR) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | From enrollment until disease progression or death (whichever occurs first), up to approximately 36 months
  TTR is defined as the time from the date of enrollment to the first documentation of objective tumor response (CR or PR) based on RECIST v.1.1. TTR will be assessed by BICR and investigator.
Percentage of Participants With Objective Response Rate (ORR) Based on Investigator Assessment Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | Up to approximately 36 months
  ORR was the defined as the percentage of participants who achieved a best overall response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), assessed by investigator based on RECIST version 1.1. For all target, non-target, and new lesions, CR was defined as a disappearance of all lesions and PR was defined as at least a 30% decrease in the sum of diameters of all lesions.
Disease Control Rate (DCR) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | Up to approximately 36 months
  DCR is defined as percentage of participants with BOR of CR, PR, or stable disease, according to RECIST v1.1.
Maximum Plasma Concentration (Cmax) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | Cycle 1: Predose, end of infusion (EOI), 3, 6, & 24 hours post start of infusion (SOI), Days 4, 8, 15, & 22; Cycle 2: Predose & EOI; Cycle 3: Predose, EOI, 3 & 6 hours post SOI; Cycle 4, 5 & every 2 cycles up to 36 months: Predose (each cycle is 21 days)
  Cmax will be calculated using noncompartmental methods. Cmax will be assessed for I-DXd, total anti-B7-H3 antibody, and MAAA-1181a.
Time to Reach Maximum Serum Concentration (Tmax) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | Cycle 1: Predose, end of infusion (EOI), 3, 6, & 24 hours post start of infusion (SOI), Days 4, 8, 15, & 22; Cycle 2: Predose & EOI; Cycle 3: Predose, EOI, 3 & 6 hours post SOI; Cycle 4, 5 & every 2 cycles up to 36 months: Predose (each cycle is 21 days)
  Tmax will be calculated using noncompartmental methods. Tmax will be assessed for I-DXd, total anti-B7-H3 antibody, and MAAA-1181a.
Minimum Observed Concentration (Ctrough) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | Cycle 1: Predose, end of infusion (EOI), 3, 6, & 24 hours post start of infusion (SOI), Days 4, 8, 15, & 22; Cycle 2: Predose & EOI; Cycle 3: Predose, EOI, 3 & 6 hours post SOI; Cycle 4, 5 & every 2 cycles up to 36 months: Predose (each cycle is 21 days)
  Ctrough will be calculated using noncompartmental methods. Ctrough will be assessed for I-DXd, total anti-B7-H3 antibody, and MAAA-1181a.
Area Under the Curve (AUC) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | Cycle 1: Predose, end of infusion (EOI), 3, 6, & 24 hours post start of infusion (SOI), Days 4, 8, 15, & 22; Cycle 2: Predose & EOI; Cycle 3: Predose, EOI, 3 & 6 hours post SOI; Cycle 4, 5 & every 2 cycles up to 36 months: Predose (each cycle is 21 days)
  AUC will be calculated using noncompartmental methods. AUC will be assessed for I-DXd, total anti-B7-H3 antibody, and MAAA-1181a.
Terminal Half-Life (T1/2) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | Cycle 1: Predose, end of infusion (EOI), 3, 6, & 24 hours post start of infusion (SOI), Days 4, 8, 15, & 22; Cycle 2: Predose & EOI; Cycle 3: Predose, EOI, 3 & 6 hours post SOI; Cycle 4, 5 & every 2 cycles up to 36 months: Predose (each cycle is 21 days)
  T1/2 will be calculated using noncompartmental methods. T1/2 will be assessed for I-DXd, total anti-B7-H3 antibody, and MAAA-1181a.
Percentage of Participants Who Have Treatment-Emergent Antidrug Antibodies (ADA) Following Treatment With I-DXd in Participants With Pretreated ES-SCLC | Cycle 1, Cycle 2, Cycle 3 and Cycle 4 Day 1: Predose; Cycle 5 Day 1 & every 2 cycles thereafter up to approximately 36 months: Predose; End of Termination Visit; 40-day Follow-up Visit (each cycle is 21 days)
  The immunogenicity of I-DXd will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (58):
- United States (16):
  - Highlands Oncology Group, Springdale, Arkansas
  - The Cancer Specialists, Llc, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Faeber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack Meridian Health-Southern Ocean Medical Center, Manahawkin, New Jersey
  - Memorial Sloan-Kettering Cancer Center (Mskcc) - New York, New York, New York
  - Montefiore Medical Center Prime, The Bronx, New York
  - Duke University Health System, Durham, North Carolina
  - Sarah Cannon (Tennessee Oncology - Nashville), Nashville, Tennessee
  - Millennium Physicians Association, Llp, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
- China (8):
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Guangdong Provincial People'S Hospital, Guangdong
  - Zhejiang Cancer Hospital, Hangzhou
  - Linyi Cancer Hospital, Linyi
  - Fudan University Shanghai Cancer Center, Shanghai
  - Union Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan
- France (7):
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Leon Berard, Lyon
  - Hôpital Nord - Chu Marseille, Marseille
  - CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - Hopital Arnaud de Villeneuve, Montpellier
  - Institut Curie - Site de Paris, Paris
  - Hopital Tenon, Paris
- Germany (2):
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitaetsklinikum Essen, Essen
- Japan (7):
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of Jfcr, Kōtoku
  - Shizuoka Cancer Center, Nagaizumi-chō
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Ōsaka-sayama
  - Kanagawa Cancer Center, Yokohama
- South Korea (5):
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (7):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Vall Dhebron, Barcelona
  - Ico L'Hospitalet - Hospital Duran I Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario Malaga, Málaga
  - Hospital Virgen Macarena, Seville
- Taiwan (6):
  - Chang Gung Medical Foundation - Kaohsiung Branch, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital Nckuh, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Rudin CM, Johnson ML, Paz-Ares L, Nishio M, Hann CL, Girard N, Rocha P, Hayashi H, Sakai T, Kim YJ, Hu H, Qian M, Singh J, Godard J, Tang M, Ahn MJ. Ifinatamab Deruxtecan in Patients With Extensive-Stage Small Cell Lung Cancer: Primary Analysis of the Phase II IDeate-Lung01 Trial. J Clin Oncol. 2026 Feb;44(4):261-273. doi: 10.1200/JCO-25-02142. Epub 2025 Oct 14. PMID 41086386